CLINICAL TRIAL: NCT05267301
Title: Open Label Post-market Evaluation of Orally Dosed AlmegaPL on Cholesterol and Cardio-metabolic Parameters.
Brief Title: AlmegaPL CV Health Open Label Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Qualitas Health (Industry)
Collaborators: Arizona State University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: ALM-CVH-22
Record Dates: First submitted 2022-02-23; First posted 2022-03-04 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Cholesterol; Triglycerides; Omega-3; Eicosapentaenoic Acid
Keywords: Microalgae; Nannochloropsis; AlmegaPL

STUDY DESIGN:
Intervention Model Description: Self elected consumers who choose to purchase this iwi EPA andiwi Heart product containing 1000-1100 mg of AlmegaPLR
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- AlmgaPL (Experimental): New consumers of iwi self-elected to start taking 2 capsules a day with 1000 mg of AlmegaPL, containing 250 mg of eicosapentaenoic acid (EPA), 150 mg polar lipids and 15 mg chlorophyll.
  Interventions: Dietary Supplement: AlmegaPL (FDA NDIN # 826)

INTERVENTIONS:
Dietary Supplement: AlmegaPL (FDA NDIN # 826) — The investigational product iwi/Cholesterol is a commercially available capsule-form herbal (algae) supplement containing Almega®PL, a Nannochloropsis algae-derived extract rich in eicosapentaenoic acid (EPA). EPA is a type of omega-3 essential fatty acid known to play a beneficial role in protection against cardiovascular disease. Iwi/Cholesterol is the only source of long chain omega-3 that does not contain the DHA that is present in other omega-3 sources (fish oil, krill oil, other algal oils). Almega®PL was registered at the Food and Drug Administration (FDA) as a New Dietary Ingredient (NDIN) in 2014.
  Other Names: iwi Algal Oil; Nannochloropsis Oil Extract

SUMMARY:
The aim of this study is to assess the effectiveness of Almega PL, a Nannochloropsis algae-derived extract rich in eicosapentaenoic acid (EPA), on improving blood markers associated with heart health of iwi customers.

DETAILED DESCRIPTION:
The investigational product iwi/Cholesterol is a commercially available capsule-form herbal (algae) supplement containing Almega®PL, a Nannochloropsis algae-derived extract rich in eicosapentaenoic acid (EPA). EPA is a type of omega-3 essential fatty acid known to play a beneficial role in protection against cardiovascular disease.The aim of this study is to assess the effectiveness of AlmegaPL on improving blood markers associated with heart health of iwi customers.The study will involve over 200 male and female new consumers of this product and monitor their blood markers during 6 months of supplementation.

ELIGIBILITY:
Inclusion Criteria:

* New iwi/AlmegaPL subscribers.

Exclusion Criteria:

* Participants that are already taking AlmegaPL.
* Participants with serious conditions including but not limited to kidney, neurological, immunological, liver and gastrointestinal disease, any heart condition or diabetes).
* Any participant attempting conception, pregnant or breastfeeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2022-05-11 (Actual); Primary Completion 2022-11-14 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Triglyceride change from baseline | From Baseline to Month 6
  Fasting triglycerides is measured using Imaware at home cardiovascular test kit

SECONDARY OUTCOMES:
Total Cholesterol change from baseline | From Baseline to Month 6
  Fasting total cholesterol is measured using Imaware at home cardiovascular test kit
VLDL-Cholesterol change from Baseline | From Baseline to Month 6
  Fasting VLDL-cholesterol is calculated using results from Imaware at home cardiovascular test kit
LDL-cholesterol change from Baseline | From Baseline to Month 6
  Fasting LDL-cholesterol is measured using Imaware at home cardiovascular test kit
HDL-cholesterol change from Baseline | From Baseline to Month 6
  Fasting HDL-cholesterol is measured using Imaware at home cardiovascular test kit
hs-CRP change from baseline | From Baseline to Month 6
  hs-CRP is measured using Imaware at home cardiovascular test kit
Fasting glucose | From Baseline to Month 6
  Fasting glucose is measured using Imaware at home cardiovascular test kit
HbA1c change from Baseline | From Baseline to Month 6
  HbA1c is measured using Imaware at home cardiovascular test kit

CONTACTS AND LOCATIONS:
Overall Officials: Eneko Ganuza Taberna, PhD, Principal Investigator — Qualitas Health; Eghogho H Etomi, MSc, Study Director — Qualitas Health; Magdalena Amezquita, MSc, Study Director — Arizona State University; Corrie Whisner, PhD, Study Chair — Arizona State University
Locations (2):
- United States (2):
  - Arizona State University, Tempe, Arizona
  - Qualitas Health, Houston, Texas

IPD SHARING:
Plan to Share IPD: No
All trial data will be shared in an aggregated form, no individual participant data will be used.

REFERENCES:
- [Background] Rao A, Briskey D, Nalley JO, Ganuza E. Omega-3 Eicosapentaenoic Acid (EPA) Rich Extract from the Microalga Nannochloropsis Decreases Cholesterol in Healthy Individuals: A Double-Blind, Randomized, Placebo-Controlled, Three-Month Supplementation Study. Nutrients. 2020 Jun 23;12(6):1869. doi: 10.3390/nu12061869. PMID 32585854
- [Derived] Ganuza E, Etomi EH, Olson M, Whisner CM. Omega-3 eicosapentaenoic polar-lipid rich extract from microalgae Nannochloropsis decreases plasma triglycerides and cholesterol in a real-world normolipidemic supplement consumer population. Front Nutr. 2024 Feb 6;11:1293909. doi: 10.3389/fnut.2024.1293909. eCollection 2024. PMID 38379539
- See also: Online shop where new subscriptions are identified — https://iwilife.com/
- See also: At home heart health test kit web portal — https://www.imaware.health/at-home-blood-test/baseline-heart-health-test
- See also: Peer reviewed article frontiers in nutrition — https://www.frontiersin.org/articles/10.3389/fnut.2024.1293909/full

DOCUMENTS (3):
  • Study Protocol (2022-03-04): https://cdn.clinicaltrials.gov/large-docs/01/NCT05267301/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-04): https://cdn.clinicaltrials.gov/large-docs/01/NCT05267301/SAP_001.pdf
  • Informed Consent Form (2022-02-07): https://cdn.clinicaltrials.gov/large-docs/01/NCT05267301/ICF_002.pdf